CLINICAL TRIAL: NCT00000305
Title: Amphetamine Cocaine Interaction Study
Brief Title: Amphetamine Cocaine Interaction Study - 2
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Original P.I. left the institution
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Texas (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NIDA-09262-2; P50DA009262 (NIH); P50-09262-2
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Cocaine-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Dextroamphetamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Dextroamphetamine

SUMMARY:
The purpose of this study is to evaluate results of d-amphetamine - cocaine (pharmacology) interaction study.

ELIGIBILITY:
Please contact site for information.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0

CONTACTS AND LOCATIONS:
Overall Officials: John Grabowski, Ph.D., Principal Investigator — University of Texas
Locations (1):
- University of Texas Health Science Center, Houston, Texas, United States